CLINICAL TRIAL: NCT01432236
Title: A Phase 3b Multicenter, Double-blind, Randomized, Placebo-controlled, 2-way Crossover Study Of Pregabalin In The Treatment Of Fibromyalgia With Concurrent Antidepressant Therapy For Comorbid Depression (Protocol A0081275)
Brief Title: A Phase 3b Multicenter Study of Pregabalin in Fibromyalgia Subjects Who Have Comorbid Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081275; 2011-002480-19 (EudraCT Number)
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2014-10

CONDITIONS: Fibromyalgia
Keywords: Pregabalin; Lyrica; depression
MeSH Terms: conditions — Fibromyalgia; Depression | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Group 1 as Pregabalin vs. Placebo (cross over study in which period one has this group)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Group 2 as placebo vs. pregabalin (cross over study in which period two will have this group)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 300 or 450 mg/day dosed BID ( twice a day) for 14 weeks; 150 mg/day starting dose
  Arms: Pregabalin
Drug: placebo — placebo capsules twice a day for 14 weeks
  Arms: Placebo

SUMMARY:
The intent of this study is to identify and treat fibromyalgia subjects with comorbid depression who are receiving an SSRI (selective serotonin reuptake inhibitor) or SNRI (selective norepinephrine reuptake inhibitor) primarily for their depression and to determine whether pregabalin demonstrates improvement relative to placebo in improving pain associated with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of any race or ethnicity who are at least 18 years of age.
* Adult women and men with a diagnosis of fibromyalgia and stable depression (major depressive disorder, depression not otherwise specified (NOS), or dysthymia) who have been taking an antidepressant (SSRI or SNRI) primarily for their depression for at least 3 months.

Exclusion Criteria:

* Have failed pregabalin treatment due to lack of improvement of symptoms at doses of greater than or equal to 300 mg daily, cannot tolerate pregabalin or any pregabalin ingredient, or participated in a pregabalin clinical trial. If the subject has taken pregabalin and discontinued for reason other than lack of improvement or intolerance, then they will be eligible. Pregabalin use within the last 30 days (prior to V1) is not permitted.
* Patients with severe or unstable depression are not eligible.
* Patients with other types of pain or conditions that may make it difficult to evaluate fibromyalgia symptoms are not eligible
* Any subject considered at risk of suicide or self harm based on investigator judgment and/or the details of a risk assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (26):
  - Genova Clinical Research, Tucson, Arizona
  - SDS Clinical Trials, Orange, California
  - Research Across America, Santa Ana, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Florida Medical Center & Research, Inc., Coral Gables, Florida
  - Meridien Research, Tampa, Florida
  - Medical Research and Health Education Foundation, Inc., Columbus, Georgia
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Social Psychiatry Research Institute, Brooklyn, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Behavioral Medicine Center, Wyomissing, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Coastal Medical, East Greenwich, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Fatigue Consultation Clinic, Salt Lake City, Utah
  - Lifetree Clinical Research, LC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
- Canada (3):
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - Canadian Centre for Clinical Trials, Thornhill, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Italy (2):
  - Azienda Ospedaliera Luigi Sacco - Polo Universitario, Milan
  - Università degli Studi di Roma "La Sapienza", Roma
- Spain (6):
  - Hospital de lˊEsperança, Barcelona
  - Instituto Universitario USP Dexeus, Barcelona
  - Servicio de Reumatologia,Institut Ferran de Reumatologia-Clinica CIMA, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital General Universitario Gregorio Marañon, Madrid

REFERENCES:
- [Derived] Bateman L, Sarzi-Puttini P, Burbridge CL, Landen JW, Masters ET, Bhadra Brown P, Scavone JM, Emir B, Vissing RS, Clair AG, Pauer LR. Burden of illness in fibromyalgia patients with comorbid depression. Clin Exp Rheumatol. 2016 Mar-Apr;34(2 Suppl 96):S106-13. Epub 2016 Mar 10. PMID 27057659
- [Derived] Arnold LM, Sarzi-Puttini P, Arsenault P, Khan T, Bhadra Brown P, Clair A, Scavone JM, Driscoll J, Landen J, Pauer L. Efficacy and Safety of Pregabalin in Patients with Fibromyalgia and Comorbid Depression Taking Concurrent Antidepressant Medication: A Randomized, Placebo-controlled Study. J Rheumatol. 2015 Jul;42(7):1237-44. doi: 10.3899/jrheum.141196. Epub 2015 Jun 1. PMID 26034150
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081275&StudyName=A%20Phase%203b%20Multicenter%20Study%20of%20Pregabalin%20in%20Fibromyalgia%20Subjects%20Who%20Have%20Comorbid%20Depression

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this double blind, crossover study, a total of 197 participants were randomized to either pregabalin/placebo or placebo/pregabalin treatment sequence. Of these, 193 took at least one dose of study medication. Four randomized participants never took study medication. Randomized participants were recruited from 4 countries at 38 study centers.
Pre-assignment Details: Participants with mean Numeric Rating Scale (NRS) pain score of ≥4 at Baseline and meeting all other inclusion/exclusion criteria were randomly assigned to receive double blind treatment with either pregabalin followed by placebo with background antidepressant or placebo followed by pregabalin with background antidepressant.
Groups:
- Pregabalin/Placebo: Participants were randomized in a 1:1 ratio to double-blind treatment with pregabalin for 6 weeks (3 weeks dose optimization and 3 weeks fixed dose) in period 1 followed by placebo in period 2 with background antidepressants. Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process. There was a 2-week single-blind taper/washout period between treatment periods.
- Placebo/Pregabalin: Participants were randomized in a 1:1 ratio to double-blind treatment with placebo for 6 weeks in period 1 followed by pregabalin in period 2 (3 weeks dose optimization and 3 weeks fixed dose) with background antidepressants. Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process. There was a 2-week single-blind taper/washout period between treatment periods.
Period: Overall Study
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Started | 96 | 97
Completed | 70 | 79
Not Completed | 26 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin | Total
Number analyzed (Participants) | 96 | 97 | 193
Age, Customized [Number; unit: Participants]
  < 18 Years | 0 | 0 | 0
  18-44 Years | 22 | 29 | 51
  45-64 Years | 69 | 60 | 129
  >= 65 Years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 93 | 180
  Male | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean NRS Pain Score at End of Period.
Description: The daily pain diary consists of an 11-point numeric scale (NRS) ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants describe their pain during the past 24 hours by choosing the appropriate number between 0 and 10. The endpoint mean pain scores for Period 1 and Period 2 are defined as the mean of the last 7 non-missing daily diary pain ratings while taking study medication in the double-blind phase during Period 1 and Period 2, respectively.
Time Frame: End of each period, at Weeks 6 and 14
Population: ITT population defined as all participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Pregabalin: The below table included participants who received pregabalin in either treatment period pooled together due to the crossover study design. This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (3 weeks dose optimization and 3 weeks fixed dose for each treatment period). Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process. There was a 2-week single-blind taper/washout period between treatment periods.
- Placebo: The below table included participants who received placebo in either treatment period pooled together due to the crossover study design. This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (3 weeks dose optimization and 3 weeks fixed dose for each treatment period). There was a 2-week single-blind taper/washout period between treatment periods.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Units on a scale | 4.84 (0.15) | 5.45 (0.16)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — Primary analysis was two-sided and performed at the 0.05 significance level; Satterthwaite's approximation was used to estimate denominator degrees of freedom; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.91 to -0.31]

2. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ) Score at Baseline.
Description: This was a 20-item participant reported outcome instrument. It contained 10 subscales, which were combined to yield a total score. The first 11 questions were related specifically to physical functioning subscale, ranging from 0 to 10. The remaining 9 questions assessed pain, fatigue, stiffness, difficulty working, and symptoms of anxiety and depression ranging from 0 to 10. The higher values indicated greater impairment. All 20 were combined to form a total score ranging from 0 to 100, provides an estimation of fibromyalgia impact with higher scores indicating more impairment. The severity categorizations for the FIQ are: less than 40 (mild), 40-60 (moderate), and above 60 (severe).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo/Pregabalin: Participants were randomized in a 1:1 ratio to double-blind treatment with placebo for 6 weeks in period 1 followed by pregabalin in period 2 (3 weeks dose optimization and 3 weeks fixed dose) with background antidepressants. Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process in period 2. There was a 2-week single-blind taper/washout period between treatment periods
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 96 | 97
Units on a scale
  Total (N=96, 96) | 63.83 (11.58) | 62.75 (12.51)
  Physical Impairment (N=96, 97) | 4.58 (2.10) | 4.44 (2.14)
  Feel Good (N=96, 97) | 7.78 (2.47) | 7.43 (2.32)
  Work Missed (N=96, 97) | 3.38 (2.88) | 3.49 (3.21)
  Do Work (N=96, 97) | 6.61 (2.03) | 6.38 (2.21)
  Pain (N=96, 96) | 6.98 (1.25) | 7.09 (1.32)
  Fatigue (N=96, 97) | 8.17 (1.37) | 8.08 (1.58)
  Rested (N=96, 97) | 7.90 (1.51) | 7.82 (1.96)
  Stiffness (N=96, 97) | 7.56 (1.76) | 7.64 (1.58)
  Anxiety (N=96, 97) | 5.65 (2.73) | 5.60 (2.59)
  Depression (N=96, 97) | 5.23 (2.64) | 4.84 (2.55)

3. Secondary Outcome: FIQ Score at End of Period.
Description: as for outcome 2
Time Frame: End of each period, at Weeks 6 and 14
Population: ITT population defined as all participants who were randomized, treated (ie, received at least one dose of study medication) and had at least one post-randomization efficacy evaluation. Different number (N) for each category represents participants that were actually treated with pregabalin and placebo during the study.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 181 | 177
Units on a scale
  Total (N=176, 172) | 43.78 (1.42) | 50.38 (1.43)
  Physical impairment (N=176, 173) | 3.35 (0.17) | 3.77 (0.17)
  Feel good (N=176, 173) | 4.69 (0.23) | 5.53 (0.23)
  Work missed (N=176 , 173) | 2.02 (0.21) | 2.62 (0.21)
  Do work (N=176, 172) | 4.56 (0.20) | 5.31 (0.20)
  Pain (N=176, 173) | 4.91 (0.17) | 5.54 (0.17)
  Fatigue (N=176, 173) | 6.32 (0.19) | 6.76 (0.19)
  Rested (N=176, 173) | 5.64 (0.19) | 6.41 (0.19)
  Stiffness (N=176, 173) | 5.24 (0.19) | 5.95 (0.19)
  Anxiety (N=176, 173) | 3.80 (0.20) | 4.35 (0.21)
  Depression (N=176, 173) | 3.20 (0.20) | 4.13 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the FIQ total score. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Analysis was conducted using a two-sided test with α=0.05. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made; Mean Difference (Final Values) = -6.60, 95% CI 2-sided [-9.33 to -3.87]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for parameter 'physical impairment'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0078, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.74 to -0.11]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'feel good'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.36 to -0.33]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis presented above for parameter 'work missed'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.01 to -0.18]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'do work'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.14 to -0.36]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'pain'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.00 to -0.28]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'fatigue'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0315, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.85 to -0.04]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'rested'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.17 to -0.35]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'stiffness'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.11 to -0.31]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'anxiety'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.93 to -0.17]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for the parameter 'depression'. Analysis was performed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.32 to -0.53]

4. Secondary Outcome: Patient Global Impression of Change (PGIC) at the End of Period 1.
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: End of Period 1 at Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Pregabalin: This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (3 weeks dose optimization and 3 weeks fixed dose for each treatment period). Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process. There was a 2-week single-blind taper/washout period between treatment periods.
- Placebo: This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (3 weeks dose optimization and 3 weeks fixed dose for each treatment period). There was a 2-week single-blind taper/washout period between treatment periods.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 93 | 93
Percentage of participants
  Very much improved | 10.8 | 4.3
  Much improved | 35.5 | 25.8
  Minimally improved | 28.0 | 40.9
  No change | 17.2 | 21.5
  Minimally worse | 4.3 | 6.5
  Much worse | 3.2 | 1.1
  Very much worse | 1.1 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; The PGIC variable was analyzed using Cochran Mantel-Haenszel (CMH) test with modified ridit transformation; Test type: Superiority or Other; p = 0.0637, Cochran-Mantel-Haenszel — This analysis was conducted using a two-sided test with α=0.05. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made

5. Other Pre Specified Outcome: PGIC at the End of Period 2.
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Because of the crossover design and PGIC recall period (since starting study medication), the Period 1 PGIC data were felt to provide the clearest comparison across treatments, whereas Period 2 PGIC data were felt to have a more complex interpretation. Thus PGIC at End of Period 2 was separately analyzed from PGIC at End of Period 1.
Time Frame: End of Period 2 at Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period (3 weeks dose optimization and 3 weeks fixed dose for each treatment period). Pregabalin was administered as immediate release (IR) capsule with a starting dose of 150 mg/day and increased up to 300 - 450 mg/day during the dose optimization process. There was a 2-week single-blind taper/washout period between treatment periods.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of Participants
  Very much improved | 18.3 | 8.6
  Much improved | 34.1 | 25.9
  Minimally improved | 28.0 | 38.3
  No change | 11.0 | 14.8
  Minimally worse | 6.1 | 8.6
  Much worse | 1.2 | 2.5
  Very much worse | 1.2 | 1.2
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; The PGIC variable was analyzed using CMH test with modified ridit transformation; Test type: Superiority or Other; p = 0.1160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants With >=30% and >=50% Pain Reduction Based on Daily Pain Diary.
Description: Participant with at least a 30% reduction in mean pain score from baseline (at randomization) to the endpoint at the end of each period (Visits 6 and 12) is considered a 30% responder, for the respective period. Similarly, a subject with at least a 50% reduction in mean pain score from baseline (at randomization) to the endpoint at the end of each period (Visits 6 and 12) is considered a 50% responder, for the respective period.
Time Frame: Visits 2, 6, and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Percentage of participants
  30% Responders | 45.3 | 27.7
  50% Responders | 26.0 | 15.8
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for 30% responders. Analysis was conducted using a logistic regression model using sequence, period, and treatment as fixed factors and participant within sequence and within participant error as random factors. Logit link transformation was used for the model; Test type: Superiority or Other; p = 0.0007, Regression, Logistic — This secondary analyses was conducted using a two-sided test with α=0.05. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis presented above is for 50% responders. Analysis was conducted using a logistic regression model using sequence, period, and treatment as fixed factors and participant within sequence and within participant error as random factors. Logit link transformation was used for the model; Test type: Superiority or Other; p = 0.0205, Regression, Logistic — [p-value comment as in outcome 6, analysis 1]

7. Secondary Outcome: Subjective Sleep Questionnaire - Mean Sleep Quality at End of Period.
Description: Subjective Sleep Questionnaire included 5 items: participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (NRS) for the previous night. Subjective rating of quality of sleep during the past night was done by selecting a number between 0 (very poor) and 10 (excellent). Mean sleep quality was calculated as the mean of the last seven days, the potential range of responses was therefore 0-10.
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Units on a scale | 6.15 (0.14) | 5.57 (0.14)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analyzed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-subject error as random factors; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This was done using a two-sided test with α=0.05. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [0.31 to 0.84]

8. Secondary Outcome: Subjective Sleep Questionnaire - Mean Subjective Wake After Sleep Onset at End of Period.
Description: Subjective Sleep Questionnaire included, participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (numeric rating scale) for the previous night. Subjective wake after sleep onset was the subjective estimate of the total amount of time the participant was awake after initial sleep onset until final awakening.
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Minutes | 33.38 (2.73) | 41.18 (2.76)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analyzed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -7.81, 95% CI 2-sided [-12.66 to -2.96]

9. Secondary Outcome: Subjective Sleep Questionnaire - Mean Latency to Sleep Onset at End of Period.
Description: Subjective Sleep Questionnaire included, participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (numeric rating scale) for the previous night. Subjective latency to sleep onset was the subjective estimate of the amount of time to fall asleep after lights out.
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Minutes | 33.54 (2.68) | 39.33 (2.71)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -5.80, 95% CI 2-sided [-10.29 to -1.31]

10. Secondary Outcome: Subjective Sleep Questionnaire - Mean Subjective Total Sleep Time at End of Period.
Description: Subjective Sleep Questionnaire included, participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (numeric rating scale) for the previous night. Subjective total sleep time was the subjective estimate of the total amount of time the participant was asleep after lights out until final awakening.
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Minutes | 422.98 (5.42) | 414.63 (5.48)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0511, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [-0.04 to 16.74]

11. Secondary Outcome: Subjective Sleep Questionnaire - Parameter Estimates for Subjective Number of Awakenings Per Night After Sleep Onset at End of Period.
Description: Subjective Sleep Questionnaire included, participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (numeric rating scale) for the previous night. Subjective number of awakenings after sleep onset was the subjective estimate of the total number of times the participant awakened during the night until final awakening.
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of times awakened
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 179 | 173
Number of times awakened | 0.48 (0.07) | 0.61 (0.07)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analyzed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors. Analyzed as a count variable using a generalized linear model assuming a Poisson distribution and utilizing a log link transformation; Test type: Superiority or Other; p = 0.1139, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.29 to 0.03]

12. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) at Baseline.
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A (anxiety) assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D (depression) assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 96 | 97
Units on a scale
  HADS-A (anxiety) | 8.67 (3.95) | 7.97 (3.77)
  HADS-D (depression) | 8.34 (3.59) | 7.73 (3.64)

13. Secondary Outcome: HADS at End of Period.
Description: as for outcome 12
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 176 | 173
Units on a scale
  HADS-A (anxiety) | 6.01 (0.28) | 6.96 (0.28)
  HADS-D (depression) | 6.17 (0.31) | 7.05 (0.31)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis presented in the above table is for HADS-A (anxiety). Analyzed using a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Two-sided test with α=0.05 was used. No corrections to alpha to control for potential inflation of Type I error resulting from multiple comparisons were made; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.40 to -0.50]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Analysis presented in the above table is for HADS-D (depression). Analyzed using a linear mixed effects model including sequence, period, and treatment as fixed factors and subject within sequence and within-subject error as random factors; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.37 to -0.39]

14. Secondary Outcome: Mean EuroQoL 5-Dimensions (EQ-5D) Score at Baseline.
Description: EQ-5D is a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a single index value characterizing current health status using a 100-point visual analog scale (0=worst, 100=best). EQ-5D summary index is obtained with a formula that weights each level of the dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 96 | 97
Units on a scale | 0.40 (0.31) | 0.37 (0.33)

15. Secondary Outcome: EQ-5D Score at End of Period.
Description: as for outcome 14
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 176 | 172
Units on a scale | 0.58 (0.02) | 0.56 (0.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.3854, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.06]

16. Other Pre Specified Outcome: Mean Patient Static Global Assessment (PSGA) Score at Baseline.
Description: PSGA was a single-item self-rated instrument that measured the participant's overall status on an 11-point NRS ranging from 0 (very poor) to 10 (very good).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 96 | 97
Units on a scale | 4.35 (2.04) | 4.46 (1.92)

17. Other Pre Specified Outcome: Mean PSGA Score at End of Period.
Description: PSGA was a single-item self-rated instrument that measured the participant's overall status on an 11-point numeric rating scale (NRS) ranging from 0 (very poor) to 10 (very good).
Time Frame: End of each period, at Weeks 6 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 176 | 172
Units on a scale | 5.83 (0.17) | 5.27 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0085, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [0.14 to 0.97]

18. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS) at Baseline.
Description: C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7) ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 96 | 97
Participants
  Wish to be Dead | 3 | 1
  Non-Specific Thoughts | 0 | 1
  Without Intent to Act | 0 | 0
  Some Intent to Act | 0 | 0
  Specific Plan and Intent | 0 | 0
  Actual Attempt | 0 | 0
  Non-Suicidal Self-Injurious Behavior | 0 | 0
  Interrupted Attempt | 0 | 0
  Aborted Attempt | 0 | 0
  Preparatory Acts or Behavior | 0 | 0
  Suicidal Behavior Present | 0 | 0
  Completed Suicide | 0 | 0

19. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the C-SSRS at Post-Baseline.
Description: C-SSRS assessed whether participant experienced following:completed suicide (1), suicide attempt (2) (response of Yes on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) (Yes on "preparatory acts or behavior"), suicidal ideation (4) (Yes on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7) (Yes on "Has subject engaged in non-suicidal self-injurious behavior"). Below table indicated one participant (10141023) treated with Pregabalin reported preparatory act. However upon study unblinding it was clarified that preparatory act occurred while the participant was taking placebo. Since preparatory act was reported at first visit of Period 2, by convention statistical summaries classified this under Pregabalin treatment.
Time Frame: From Visit 3 to Visit 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 181 | 177
Participants
  Wish to be Dead | 10 | 8
  Non-Specific Thoughts | 3 | 1
  Without Intent to Act | 2 | 0
  Some Intent to Act | 0 | 0
  Specific Plan and Intent | 0 | 0
  Actual Attempt | 0 | 0
  Non-Suicidal Self-Injurious Behavior | 0 | 0
  Interrupted Attempt | 0 | 0
  Aborted Attempt | 0 | 0
  Preparatory Acts or Behavior | 1 | 0
  Suicidal Behavior Present | 1 | 0
  Completed Suicide | 0 | 0

20. Other Pre Specified Outcome: Work Productivity and Activity Index-Specific Health Problem (WPAI-SHP) Questionnaire at Baseline.
Description: WPAI-SHP assessed work productivity and impairment. It was a participant-rated, six-item questionnaire regarding current employment, hours missed and actually worked, and degree to which a specified health problem affected work productivity and regular activities over the past 7 days. Subscale scores included percent work time missed due to the health problem; percent impairment while working due to problem; percent overall work impairment due to problem; and percent activity impairment due to problem. Each subscale score was expressed as an impairment percentage (0-100) where higher numbers indicated greater impairment and less productivity.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- All Participants: All randomized participants were included in this analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 193
Units on a scale
  Percent Absenteeism (N= 86) | 15.22 (25.36)
  Percent Presenteeism (N= 83) | 53.98 (21.52)
  Percent Overall Work Impairment (N= 82) | 57.96 (23.42)
  Percent Activity Impairment (N=193) | 64.97 (18.77)

21. Other Pre Specified Outcome: Health Utilization Assessment (Total Office Visits, Number of Hospitalizations and Number of Emergency Room Visits) at Baseline.
Description: The healthcare utilization assessment was used to capture healthcare utilization data at Baseline. This assessment contained 10 questions related to aspects of healthcare services.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | All Participants
Number analyzed (Participants) | 193
Visits
  Total office visits (N= 193) | 5.01 (6.6)
  Number of hospitalizations (N= 0) | NA (NA) — Could not be calculated as N=0
  Number of emergency room visits (N= 12) | 1.83 (1.0)

22. Other Pre Specified Outcome: Health Utilization Assessment (Time for Help no Payment) at Baseline.
Description: The healthcare utilization assessment was used to capture healthcare utilization data at Baseline. This assessment contained 10 questions related to aspects of healthcare services. 'Time for help no payment' refers to time other people spent without receiving payment to help with activities the patient cannot perform due to fibromyalgia.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | All Participants
Number analyzed (Participants) | 193
Hours | 50.37 (98.1)

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/181 | 1/177
Other Adverse Events (participants affected / at risk) | 139/181 | 106/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=181) | Placebo (N=177)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Detoxification (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=181) | Placebo (N=177)
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 3 | 0
Eye disorder (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 7 | 3
Visual impairment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 19 | 4
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 7
Dry mouth (Gastrointestinal disorders) | 12 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 12
Odynophagia (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 3 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 2
Crying (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Energy increased (General disorders) | 1 | 0
Fatigue (General disorders) | 12 | 8
Feeling abnormal (General disorders) | 5 | 0
Feeling drunk (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Feeling jittery (General disorders) | 2 | 0
Gait disturbance (General disorders) | 3 | 0
Hunger (General disorders) | 3 | 1
Inflammation (General disorders) | 1 | 0
Irritability (General disorders) | 3 | 1
Malaise (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 7 | 3
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 4
Swelling (General disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2
Bronchitis viral (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 2
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 4 | 2
Influenza (Infections and infestations) | 3 | 2
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 10
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 3 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 3
Eosinophil count increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 16 | 3
Fluid retention (Metabolism and nutrition disorders) | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Food craving (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 4 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Areflexia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 5 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Clumsiness (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 5 | 4
Dizziness (Nervous system disorders) | 51 | 12
Dizziness postural (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 14 | 17
Hypersomnia (Nervous system disorders) | 3 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 5 | 1
Mental impairment (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 3
Myoclonus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Repetitive speech (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 4 | 2
Somnolence (Nervous system disorders) | 36 | 8
Stupor (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 8 | 7
Apathy (Psychiatric disorders) | 0 | 1
Bradyphrenia (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 5 | 4
Disorientation (Psychiatric disorders) | 5 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 13 | 1
Nervousness (Psychiatric disorders) | 3 | 2
Nightmare (Psychiatric disorders) | 1 | 4
Panic attack (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Thinking abnormal (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.